CLINICAL TRIAL: NCT00487552
Title: Endoscopic Gastroenteric Anastomosis Formed by Magnetic Compression and Stent Placement for Palliation of Malignant Gastric Outlet Obstruction
Brief Title: Magnetic Anastomosis Device Relief of Malignant Gastric Outlet Obstruction
Acronym: MAD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to achieve one of the primary endpoints.
Sponsor: Cook Group Incorporated (Industry)
Collaborators: MED Institute, Incorporated (Industry); Cook Endoscopy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 06-014; 900000
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Results first posted 2012-07-27 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-07

CONDITIONS: Gastric Outlet Obstruction
Keywords: endoscopy; esophagogastroduodenoscopy; gastric outlet obstruction; gastro-jejunostomy; gastric malignancy; duodenal stent; Malignant Gastric Outlet Obstruction
MeSH Terms: conditions — Gastric Outlet Obstruction; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): palliative treatment of gastric outlet obstruction
  Interventions: Device: Cook Magnetic Anastomosis Device (MAD) with Stent

INTERVENTIONS:
Device: Cook Magnetic Anastomosis Device (MAD) with Stent — Gastro-jejunal anastomosis

SUMMARY:
The purpose of this study is to determine if the Cook Magnetic Anastomosis Device can be used to safely and successfully create a patent gastrojejunal anastomosis in subjects requiring treatment of gastric outlet obstruction caused by malignancy.

DETAILED DESCRIPTION:
Surgical treatments for malignant gastric outlet obstructions carry substantial risks and are associated with postoperative morbidity. External compression from advancing tumor or tissue growth through the stent can cause stenosis or re-obstruction. In these patients, the creation of a patent fistula that allows gastric emptying may significantly improve palliation. Minimally invasive techniques that carry no greater risks than enteral stenting may provide a viable palliative treatment. The primary objectives are safety, and successful creation of a gastro-jejunal anastomosis. Secondary objectives are successful resumption or improvement in the ability to tolerate PO feeding, rate of stent migration, and duration of stent and anastomosis patency.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable malignancy with, or at risk of developing gastric outlet obstruction with GOOSS ≤ 2
* Karnofsky Performance Score ≥ 60

Exclusion Criteria:

* Patient is unable to understand and execute informed consent
* Age below 18 years
* Patients with any prior gastrointestinal surgery that significantly alters gastrojejunal anatomy
* Implanted cardiac pacemaker, defibrillator or ventricular assist device
* Requirement for chronic anticoagulation, or with uncorrectable coagulopathy
* Patients receiving chronic steroids or other drugs that may impair wound healing or formation of an intact anastomosis
* Simultaneously participating in another investigational drug or device
* Patients with suspicion of, or documented multiple small bowel strictures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Fockens, MD, PhD, Principal Investigator — Amsterdam Academic Medical Center
Locations (4):
- Hospital de Erasme, Brussels, Belgium
- Instituto di Clinical Chirurgica, Rome, Italy
- Netherlands (2):
  - Amsterdam Academic Medical Center, Amsterdam
  - University Medical Center Utrecht, Utrecht

RESULTS

PARTICIPANT FLOW:
Groups:
- Magnetic Anastomosis Device (MAD) With Stent: Magnetic Anastomosis Device used with gastro-jejunal or duodenal stent for palliative treatment of gastric outlet obstruction.
Period: Overall Study
Arm/Group | Magnetic Anastomosis Device (MAD) With Stent
Started | 18
Completed | 12
Not Completed | 6
Not completed — Unsuccessful magnet placements | 3
Not completed — Death due to progressive malignancy | 2
Not completed — Stent not placed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Magnetic Anastomosis Device (MAD) With Stent
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 13
Karnofsky Score [Mean (Standard Deviation); unit: Units on a scale] — The Karnofsky score allows patients to be classified as to their functional impairment. It runs from 100 to 0, where 100 is "perfect" health and 0 is death.
  Units on a scale | 72.2 (9.4)
Presenting Condition [Number; unit: participants]
  Cholangio cancer | 3
  Gastric cancer | 1
  Pancreatic cancer | 12
  Other | 2
Current Treatments [Number; unit: participants]
  Chemotherapy | 4
  Radiotherapy | 0
  Brachytherapy | 0
  No treatment - Palliative care only | 10
  Other | 1
  Patients with no current treatments | 3

OUTCOME MEASURES:

1. Primary Outcome: Success Rate Associated With the Creation of a Gastro-jejunal Anastomosis Using the Cook Magnetic Anastomosis Device With Trans-anastomotic Deployment of a Gastro-jejunal or Duodenal Stent
Description: Success is defined as placement of the gastric and jejunal magnets, creation of the anastomosis, and deployment of the gastro-jejunal stent.
Time Frame: Approximately 8-10 days
Measure: Number; unit: participants
Arm/Group | Magnetic Anastomosis Device (MAD) With Stent
Number analyzed (Participants) | 18
participants | 12

2. Post Hoc Outcome: Success Rate of Mature Anastomosis Creation Using Magnetic Anastomosis Device (MAD)
Description: Endoscopy was performed to determine whether an anastomosis (hole) was successfully created.
Time Frame: Approximately 8-10 days
Population: Patients who underwent a second endoscopy after successful magnet placement
Measure: Number; unit: participants
Groups:
- Magnetic Anastomosis Device (MAD): Magnetic Anastomosis Device (MAD) used for palliative treatment of gastric outlet obstruction.
Arm/Group | Magnetic Anastomosis Device (MAD)
Number analyzed (Participants) | 13
participants | 13

ADVERSE EVENTS:
Description: Only 12 of 18 patients are reported in the reported Adverse Events section as "Total Number of Participants at Risk". These are the participants that received both the magnets and the stent (primary success).
Arm/Group | Magnetic Anastomosis Device (MAD) With Stent
Serious Adverse Events (participants affected / at risk) | 10/12
Other Adverse Events (participants affected / at risk) | 4/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnetic Anastomosis Device (MAD) With Stent (N=12)
Death (Blood and lymphatic system disorders) | 1 (1) — Death was due to peritonitis/sepsis subsequent to stent migration.
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) — Deaths were due to progressive malignancy.
Death (Cardiac disorders) | 1 (1) — Death was due to co-morbidity.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnetic Anastomosis Device (MAD) With Stent (N=12)
Migration (Gastrointestinal disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
Enrollment was stopped in Feb 2009, due to the death of a patient after distal stent migration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each PI/site is restricted from making any publication until the multi-center publication has been presented (published) or 12 months after conclusion/abandonment/or termination of the Study (in the case where the multi-center publication has not been submitted within the 12 months) or Cook confirms there will be no multi-center publication.